CLINICAL TRIAL: NCT01257126
Title: Efficacy of Diclofenac Potassium Versus Nimesulide in the Treatment of Fever and Pain in Children Aged 3 to 7 Years With Community Acquired, Non-complicated, Upper Respiratory Tract Infection
Brief Title: Efficacy of Diclofenac Potassium vs Nimesulide in the Treatment of Fever and Pain in Children With Upper Respiratory Tract Infection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCAT458CMX01
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Upper Respiratory Tract Infections
Keywords: Upper respiratory tract infections; diclofenac potassium; nimesulide; fever; pain
MeSH Terms: conditions — Respiratory Tract Infections; Fever; Pain | interventions — Diclofenac; nimesulide

ARMS (2):
- diclofenac potassium (Experimental)
  Interventions: Drug: diclofenac potassium
- nimesulide (Active Comparator)
  Interventions: Drug: nimesulide

INTERVENTIONS:
Drug: diclofenac potassium
  Arms: diclofenac potassium
Drug: nimesulide
  Arms: nimesulide

SUMMARY:
This is a local, phase IV, open-label, randomized, head to head study of children aged 3 to 7 years. The objective of the study is to compare the efficacy of a single dose of both diclofenac potassium and nimesulide in the reduction of fever and pain secondary to upper respiratory tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Children who present community acquired, non-complicated, upper respiratory tract infection: rhino-sinusitis, pharyngitis, tonsillitis, ear infection or the combination of these.
* Child must present axillary temperature ≥ 37.5°C.

Exclusion Criteria:

* Prior history of allergic reaction to the components of the study medication.
* Use of any NSAID or pharmacologic agent in the 24 hours prior to visit 1.
* Subjects who, in the opinion of the investigator, have developed, or are at risk of developing, a complicated infection and are not suitable subjects for the purposes of the study.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of fever as measured by axillary temperature | 120 minutes

SECONDARY OUTCOMES:
Reduction of pain as measured by visual analog scale | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals